CLINICAL TRIAL: NCT07106242
Title: Japan Post Market Adaptive Deep Brain Stimulation (aDBS) Study (Early Adapter) Part II
Brief Title: Adaptive Deep Brain Stimulation (aDBS) Study (Early Adapter) Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MDT20041
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- aDBS Preferred Mode (Experimental)
  Interventions: Device: Adaptive DBS
- cDBS (Active Comparator)
  Interventions: Device: cDBS

INTERVENTIONS:
Device: Adaptive DBS — Subjects will receive Dual or Single Threshold aDBS which are acceptable
  Arms: aDBS Preferred Mode
Device: cDBS — cDBS
  Arms: cDBS

SUMMARY:
The purpose of the study is to evaluate the efficacy of aDBS (preferred mode, single or dual threshold) vs standard continuous DBS (cDBS) in decreasing Total Electrical Energy Delivered (TEED). Prospective randomized, single-blind, crossover, multicenter study of aDBS in subjects with Parkinson's disease.

DETAILED DESCRIPTION:
Prospective randomized, single-blind, crossover, multicenter study of aDBS in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Parkinson's disease with motor impairments.
2. Subject is implanted with Percept PC and Medtronic DBS leads and extensions bilaterally in the same target (physician confirmed), STN or GPi.
3. Subject has completed Early Adapter 1 study OR if the subject has not completed Early Adapter 1, she/he has documented evidence that aDBS is well tolerated in at least one mode (single or dual threshold) (Note: Tolerance means that the investigator has determined that aDBS is suitable for PD treatment). For subject who only tolerated dual threshold mode, aDBS must be set up in both hemispheres.
4. Subject has Beta band (8-30 Hz) amplitude ≥ 1.2 μVp detected on either left and/or right DBS leads on sensing channels 0-2, 0-3, or 1-3; 8-10, 8-11, or 9-11; As assessed in screening from Early Adapter I study. For subjects who have not completed Early Adapter Part I, it can be assessed using the record of standard test of eligibility for aDBS at the site.
5. The subject responds to DBS Therapy.
6. The subject's cDBS parameters and PD medications are stable and expected to remain stable from enrollment through the end of the aDBS treatment phase. (Note: Stability is defined as no major changes in cDBS parameter and medication for the last 30 days prior to aDBS setup or as defined by the physician.)
7. Subject is configured to monopolar or dual monopolar stimulation using contacts 1 and/or 2 (9 and/or 10) on at least one side
8. Subject is willing and able to attend all study-required visits and complete the study procedures.
9. Subject has the ability to understand and provide written informed consent for participation in the study prior to the study-related procedures being conducted.
10. Subject is a male or non-pregnant female. If female of childbearing potential, and if sexually active, must be using, or agree to use, a medically acceptable method of birth control as confirmed by the investigator.

Exclusion Criteria:

1. Subject and/or caregiver is unable to utilize the patient programmer.
2. Subject has more than one lead in each hemisphere of the brain.
3. Subject has cortical leads or additional unapproved hardware implanted in the brain.
4. Subject has more than one INS.
5. No tested mode of aDBS (single or dual threshold) is tolerated. (Note: Tolerance is defined that investigator has determined that aDBS is suitable for PD treatment.).
6. At enrollment, the subject's INS has a predicted battery life of <1 year.
7. Subject has untreated severe depression which may preclude them from study participation.
8. Subject requires diathermy, transcranial magnetic stimulation (TMS), electroconvulsive therapy (ECT), or Magnetic resonance-guided focused ultrasound (MRgFUS).
9. Subject has a metallic implant in the head, (e.g., aneurysm clip, cochlear implant).
10. Subject has, or plans to obtain, an implanted electrical stimulation medical device anywhere in the body (e.g., cardiac pacemaker, defibrillator, spinal cord stimulator).
11. Subject has, or plans to obtain, an implanted medication pump for the treatment of Parkinson's disease (e.g., CADD-Legacy1400 pump) and/or portable infusion pump.
12. The subject has an abnormal neurological examination that would preclude him from study participation.
13. Subject is breast feeding.
14. Subject is under the age of 20 years.
15. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study.
16. Subjects with signal artifact on all 6 aDBS sense pathways (3 on each of both DBS leads) which preclude the clinician from setting thresholds* *As assessed in aDBS setup from Early Adapter Part I and aDBS data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Total Electrical Energy Delivered (TEED) during adaptive (aDBS) as compared to continuous DBS (cDBS) | A 45-day period of aDBS treatment will be compared to a 45-day period of cDBS treatment

SECONDARY OUTCOMES:
The mean percent time within an optimal beta LFP threshold of beta LFP power during aDBS mode compared to cDBS | A 45-day period of aDBS treatment will be compared to a 45-day period of cDBS treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Juntendo University Nerima Hospital, Tokyo, Nerima-ku
  - Juntendo University Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No